CLINICAL TRIAL: NCT04128085
Title: A Phase I, Open-label, Multicenter, Dose Escalation and Expansion Study to Evaluate the Tolerance and Pharmacokinetics of TQB3804 in Subjects With Advanced Malignant Tumors
Brief Title: A Study to Evaluate the Tolerance and Pharmacokinetics of TQB3804 in Subjects With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3804-I-01
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3804 (Experimental): TQB3804 tablet administered orally , once daily in 28-day cycle.
  Interventions: Drug: TQB3804

INTERVENTIONS:
Drug: TQB3804 — A kind of tyrosine kinase inhibitor.

SUMMARY:
This is a study to evaluate the tolerance, dose-limiting toxicity (DLT), phase II recommended dose (RP2D), and maximum tolerated dose (MTD) of single and multiple oral doses of TQB3804 in patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

- 1. Understood and signed an informed consent form. 2. 18 and 70 years old. 3. Histologically or cytologically confirmed advanced malignant tumor. 4. Has EGFR mutations. 5. Life expectancy ≥12 weeks. 6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2.

7.Adequate organ system function. 8.At least one measurable lesion.

Exclusion Criteria:

* 1.Hypersensitivity to TQB3804 or its excipient. 2. Has diagnosed and/or treated additional malignancy within 5 years with the exception of cured carcinoma in situ of the cervix、intramucosal carcinoma of gastrointestinal tract、breast and non-melanoma skin cancers and superficial bladder tumors.

  3.Has interstitial pneumonia. 4.Brain metastases with symptom . 5.Has currently uncontrollable congestive heart failure. 6.Has history of arterial thromboembolism within 6 months. 7.Has any bleeding tendency or coagulopathy within 6 months. 8.Has skin toxicity ≥ grade 2 within 4 weeks. 9.Has serious gastrointestinal diseases within 4 weeks. 10.Has received any major surgery within 4 weeks. 11.Participated in other clinical trials within 4 weeks. 12.Has active viral, bacterial and fungal infections within 4 weeks. 13.Has received any cancer therapy within 4 weeks or 5 times of t1/2. 14.Has ≥ grade 2 toxicity caused by previous anti-tumor treatment. 15. HBsAg positive and HBV DNA positive (≥ULN);HCV antibody and HCV-RNA positive (≥ULN); HIV positive or ≥HIV ULN.

  16. Has multiple factors affecting oral medication. 17. Breastfeeding or pregnant women.; Men unwilling to use adequate contraceptive measures during the study.

  18. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days
  Subjects appear the following toxic reaction relate to the drug after treatment within 28 days ：III °or above of non-hematological toxicity, IV° hematological toxicity , neutropenia associated with fever.

SECONDARY OUTCOMES:
Cmax | Hour 0, 1, 2, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 168 hours post-dose on single dose; Hour 0 of day 8,day 15,day14,day 22,day 28 on multiple dose and Hour 0, 1, 2, 4, 6, 8, 10, 12, 18, 24 hours post-dose on multiple dose of day 28.
  Cmax is the maximum plasma concentration of TQB3804 or metabolite(s).
Tmax | Hour 0, 1, 2, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 168 hours post-dose on single dose; Hour 0 of day 8,day 15,day14,day 22,day 28 on multiple dose and Hour 0, 1, 2, 4, 6, 8, 10, 12, 18, 24 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3804 by assessment of time to reach maximum plasma concentration.
AUC0-t | Hour 0, 1, 2, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 168 hours post-dose on single dose; Hour 0 of day 8,day 15,day14,day 22,day 28 on multiple dose and Hour 0, 1, 2, 4, 6, 8, 10, 12, 18, 24 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3804 by assessment of area under the plasma concentration time curve from zero to infinity.
Progression Free Survival (PFS) | Baseline up to 52 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Objective Response Rate(ORR) | Baseline up to 52 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease Control Rate(DCR) | Baseline up to 52 weeks
  Percentage of participants achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China